CLINICAL TRIAL: NCT01222221
Title: A Cancer Research UK Phase I Trial of IMA950 (A Novel Multi-Peptide Vaccine) Plus GM-CSF in Patients With Newly Diagnosed Glioblastoma
Brief Title: Vaccine Therapy, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000686559; CRUK-CR0902-11; EUDRACT-2009-015971-28
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult gliosarcoma; adult giant cell glioblastoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Gliosarcoma; Glioblastoma | interventions — IMA950; sargramostim; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Biological: glioblastoma multiforme multipeptide vaccine IMA950
Biological: sargramostim
Drug: temozolomide
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving vaccine therapy together with temozolomide and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy when given together with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety and tolerability of glioblastoma multiform multi-antigen vaccine IMA950 plus sargramostim (GM-CSF) in combination with standard chemoradiotherapy comprising temozolomide and radiotherapy followed by adjuvant temozolomide in patients with newly diagnosed glioblastoma multiforme.
* To determine the immunogenicity of this regimen in these patients.

Secondary

* To determine the anti-tumor effect of this regimen in these patients.
* To determine the effect of pre-treatment levels of regulatory T-cells on the immunogenicity of this regimen in these patients. (Exploratory)
* To evaluate the potential effect of steroid dose on the immunological response to glioblastoma multiform multi-antigen vaccine IMA950 plus GM-CSF.

Tertiary

* To assess the level of O6-methyl-DNA-methyltransferase (MGMT) promoter methylation in tumor tissue and any potential association with any observed anti-tumor effect.
* To evaluate the kinetics of the observed immunogenicity of glioblastoma multiform multi-antigen vaccine IMA950 plus GM-CSF.
* To explore the possible biomarker signatures that may predict immunological response to glioblastoma multiform multi-antigen vaccine IMA950 plus GM-CSF. (Exploratory)
* To explore the possible effects of this regimen on any observed pseudo-progression and pseudo-regression in these patients. (exploratory)

OUTLINE: This is a multicenter study. Patients are recruited to cohort 1 or 2 with priority recruitment to cohort 1. All patients undergo standard chemoradiotherapy followed by adjuvant temozolomide as planned.

* Standard therapy (chemoradiotherapy and adjuvant temozolomide): Beginning after surgery, patients receive chemoradiotherapy comprising oral temozolomide daily for 6 weeks and radiotherapy once daily, 5 days a week for 6 weeks. Beginning 35 days after completion of radiotherapy, patients receive adjuvant oral temozolomide alone on days 1-5. Treatment with temozolomide repeats every 28 days for 6 courses.
* Vaccine therapy: Patients also receive vaccine therapy beginning at one of two time points. Patients are recruited into 1 of 2 cohorts that differ in the timing of the vaccination schedule in relation to a patient's standard therapy.

  * Cohort 1: Vaccination begins 7-14 days prior to chemoradiotherapy.

    * Induction phase: Patients receive the first 6 doses of sargramostim intradermally (ID) followed by glioblastoma multiform multi-antigen vaccine IMA950 ID on days 1, 2, 3, 8, 15, and 22 in the absence of disease progression or unacceptable toxicity.
    * Maintenance phase: Patients receive sargramostim followed by glioblastoma multiform multi-antigen vaccine IMA950 ID on days 50 and 78 and then on day 21 of each adjuvant temozolomide course, beginning in course 1, for 3 courses in the absence of disease progression or unacceptable toxicity.
  * Cohort 2: Vaccination begins at least 7 days after chemoradiotherapy and 28 days prior to adjuvant temozolomide.

    * Induction phase: Patients receive the first 6 doses of sargramostim followed by glioblastoma multiform multi-antigen vaccine IMA950 ID as in cohort 1 induction phase, beginning at a different time point.
    * Maintenance phase: Patients receive sargramostim followed by glioblastoma multiform multi-antigen vaccine IMA950 ID on day 21 of each adjuvant temozolomide course, beginning in course 1, for 5 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacodynamic, biomarker, and immunologic studies.

After completion of study treatment, patients are followed at 41 weeks.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed glioblastoma multiforme (astrocytoma WHO grade IV disease)

  * Newly diagnosed disease
  * Resectable tumor (not including patients undergoing biopsy only or tumors involving the brain stem or cerebellum)
* Meets 1 of the following criteria regarding standard chemoradiotherapy:

  * Cohort 1

    * Eligible for standard chemoradiotherapy with temozolomide followed by adjuvant temozolomide

      * Has undergone surgical resection before study enrollment
  * Cohort 2

    * Completed standard chemoradiotherapy with temozolomide with no subsequent progression of disease
* Expected to complete standard chemoradiotherapy and 6 courses of adjuvant temozolomide
* HLA-A*02 positive

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 30 weeks
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Lymphocyte count ≥ 1.0 x 10^9/L (cohort 1) OR ≥ 0.35 x 10^9/L post-chemoradiotherapy and ≥ 1.0 x 10^9/L prior to the start of chemoradiotherapy (cohort 2)
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 3.0 times ULN
* Alkaline phosphatase ≤ 3.0 times ULN
* Hepatitis B serology negative (HBcAg-seronegative)
* No known hepatitis C or HIV serological positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use one (male) or two (female) highly effective forms of contraception 2 weeks before, during, and for 6 months after completion of study therapy
* Not at high medical risk due to nonmalignant systemic disease including active uncontrolled infection
* No known hypersensitivity to GM-CSF or excipients
* No history of autoimmune disease
* No concurrent congestive heart failure
* No prior history of NYHA class III-IV cardiac disease, cardiac ischemia, or cardiac arrhythmia
* No other condition that might interfere with the patient's ability to generate an immune response
* No other condition that, in the investigator's opinion, would make the patient not a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 7 days since prior dexamethasone (dose > 4 mg daily or equivalent)
* At least 4 weeks since prior major surgery for any condition (except surgical resection as part of primary standard therapy in cohort 1)
* At least 30 days since prior and no concurrent participation in another clinical trial or planning to participate in another interventional clinical trial (concurrent participation on an observational study allowed)
* At least 30 days since prior and no other concurrent investigational drugs
* No prior treatment for glioblastoma including Gliadel Wafers

  * Early components of standard therapy are allowed if already initiated (i.e., surgical resection [cohort 1] or surgical resection followed by conventional external-beam radiotherapy and concomitant temozolomide [cohort 2])
* No other concurrent anticancer therapy
* No other concurrent vaccinations from 2 weeks before the first study vaccine to the end of the sixth study vaccine (the induction phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Causality of each adverse event (AE) to glioblastoma multiform multi-antigen vaccine IMA950 and GM-CSF and AE severity according to NCI CTCAE Version 4.0
Total number of patients showing patient-individual T-cell responses against a single or multiple tumor-associated peptides (TUMAP) contained in the study vaccine IMA950 at one or more post-vaccination time points by HLA multimer analysis

SECONDARY OUTCOMES:
Progression-free survival (PSF) at 6 and 9 months post-surgery as assessed by the Macdonald criteria from conventional gadolinium-enhanced MRI and clinical assessment
Correlation between steroid levels and observed T-cell responses
Correlation between O6-methyl-DNA-methyltransferase (MGMT) promoter methylation status in tumor tissue using methylation-specific polymerase chain reaction and clinical benefit (PFS at 6 months and 9 months)
Kinetics of vaccine-induced TUMAP responses including summary descriptions of the time of onset, sustainability, and magnitude of the observed response

CONTACTS AND LOCATIONS:
Overall Officials: Roy Rampling, MD, PhD, Principal Investigator — University of Glasgow
Locations (7):
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge, England
  - UCL Cancer Institute, London, England
  - Southampton General Hospital, Southampton, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Western General Hospital, Edinburgh
  - St James' University Hospital, Leeds
  - The Christie NHS Foundation Trust, Manchester